Title page:

Title: Comparison of Clinical and Radiographic Success Between:

Mineral Trioxide Aggregate (MTA) & Ferric Sulfate (FS) Pulpotomies for Primary Molars.

NCT 02783911

Date: Sep 02, 2014

## Comparison of Mineral Trioxide Aggregate and Ferric Sulfate:

## Pulpal Medicaments for Pulpotomized Primary Teeth

## Statistical analysis plan

The following clinical information were collected from the charts: Mobility, pain, abscess/draining fistula, and facial swelling. Exfoliation of the pulp treated teeth was recorded and graded as normal, early, or delayed based on the age of the patient at the time of the recall and on the exfoliation status of the contralateral tooth. If there is any clinical signs of the above the tooth will be count as clinical failure.

Data was analyzed using the Statistical Package for Social Sciences v 16.0 (SPSS Inc., Chicago, Ill). The difference between the materials was analyzed using chi-square, Significance level was set P < .05.

## **Chi-Square Tests**

| | | | Asymptotic Significance (2- | Exact Sig. (2- | Exact Sig. (1- |
|---|---|---|---|---|---|
| | Value | df | sided) | sided) | sided) |
| Pearson Chi-Square | .059ª | 1 | <mark>.808</mark> . | | |
| Continuity Correction <sup>b</sup> | .000 | 1 | 1.000 | | |
| Likelihood Ratio | .060 | 1 | .807 | | |
| Fisher's Exact Test | | | | 1.000 | .603 |
| Linear-by-Linear Association | .057 | 1 | .812 | | |
| N of Valid Cases | 24 | | | | |

a. 2 cells (50.0%) have expected count less than 5. The minimum expected count is 2.25.

Summary: The result showed there is no statistical difference in long term clinical success between the two pulpotomy medicaments. (MTA vs FS)

b. Computed only for a 2x2 table